CLINICAL TRIAL: NCT02901834
Title: PainSquad+: A Smartphone App to Support Real-time Pain Management for Adolescents
Brief Title: PainSquad+: A Smartphone App to Support Real-time Pain Management for Adolescents With Cancer
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 100045124
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Therapy-Associated Cancer
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Adolescents with cancer (AWC) are in a unique developmental stage that may mean pain characteristics, the impact of pain, and pain treatment outcomes are different in adolescents compared to children and adults. In response, we will develop and test the PainSquad+ pain management smartphone app. First, we will conduct usability testing to refine PainSquad+ so that it is useable, acceptable and understandable for AWC. Secondly we will: (a) test the feasibility of conducting a large-scale PainSquad+ experiment and (b) begin to examine how effective PainSquad+ is at helping adolescents manage pain. We hope that once developed and tested for effectiveness, PainSquad+ will improve pain treatment and ultimately quality of life in AWC.

DETAILED DESCRIPTION:
Using a conservative estimate of 7 adolescents per cycle and 3 testing cycles, 21 adolescents will take part in usability testing of the PainSquad+ prototype. Recruitment will be conducted in a single hematology/oncology division of a metropolitan and university-affiliated pediatric tertiary care center in Toronto, Canada. This site hosts one of the largest cancer programs in North America, with approximately 350 new diagnoses each year. Based on our previous research at this site, 72 ± 4% (M ± SD; range = 67-75%) of eligible AWC agreed to participate in similar studies (unpublished data). Convenience sampling will be used to recruit eligible individuals. The testing procedures will commence after eligibility is assessed, informed consent is obtained, and demographic and baseline outcome data are collected. Inclusion criteria will be: (a) aged 12-18 years, (b) able to speak and read English, (c) actively undergoing cancer treatment on an in- or out-patient basis, (d) being at least 3 months from diagnosis and (d) having self-reported pain of any intensity in the week immediately prior to recruitment. Exclusion criteria will be: (a) one or more major co-morbid (medical or psychiatric) conditions that would preclude use of a smartphone, and (b) palliative/end-of-life patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-18 years,
* able to speak and read English
* actively undergoing cancer treatment on an in- or out-patient basis
* being at least 3 months from diagnosis
* having self-reported pain of any intensity in the week immediately prior to recruitment

Exclusion Criteria:

* one or more major co-morbid (medical or psychiatric) conditions that would preclude use of a smartphone
* palliative/end-of-life patients.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents aged 12-18 years who have been diagnosed at least 2 months with cancer and have had pain in the past week.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Accrual and attrition rates | 12 months
  The Cancer Pain Management App Recruitment Log has been designed to record data related to the number of eligible adolescents per recruitment day, reasons for ineligibility, and reasons for nonparticipation. The Cancer Pain Management App Activity Log has been designed to record data on attrition (occurrence/reasons for attrition), as well as technical difficulties, adherence and outcome measure completion.
Technical difficulties | 12 months
  The occurrence and description of technical problems will be recorded on the Cancer Pain Management App Activity Log.
Acceptability | 12 months
  The Acceptability E-Scale (AES) ascertains perceptions related to how helpful, difficult, and enjoyable e-based programs are to use, how understandable questions are, and how acceptable the time invested in reporting was (Wu, Johnson, Schepp, & Berry, 2011). For the purpose of the present study, the wording of the AES will be slightly modified. Specifically, the words "computer program" will be changed to "app" and open-ended questions regarding study acceptability will be added.
Adherence | 12 months
  Measured as the percentage of pain reports received on the secure server. An RA will sign onto the server and extract data logged by AWC on Day 29 to calculate adherence (100% when 28/28 morning and evening reports are completed). These data will be recorded on the Cancer Pain Management App Activity Log.
Outcome measure feasibility | 12 months
  Measured as the percentage of completed questionnaires at baseline and study completion. An RA will sign onto the server and extract data logged by AWC on Day 29 to calculate the percentage of completed questionnaires (100% when all questionnaires are completed). These data will be recorded on the Cancer Pain Management App Activity Log.
Pain intensity | 12 months
  Measured using the pain intensity items (current pain intensity and worst, average, and least pain intensity in the previous week) of the Brief Pain Inventory (BPI). The BPI is considered the standard for clinical and research use in cancer patients (Mathias et al., 2011). Each item is rated numerically from 0-10. Individual scores on each of the 4 items may be summed and to provide a composite pain intensity score. Individual and summary scores will be used in our analyses. Validity and reliability have been well-established in adults with cancer and the intensity sub-scale has been used successfully in AWC (Ameringer, 2010).
Pain interference | 12 months
  The Patient Reported Outcomes Measurement Information System Pediatric (PROMIS) Pain Interference Short-form Scale is an 8-item scale describing how pain restricts daily activities related to physical, psychological, and social functioning, as well as sleep, school, and enjoyment of life. Each item is scored on a 5-point Likert response scale and totaling the scores generates a summary score, which will be used in our analyses. Construct validity has been established in AWC (Hinds et al., 2013).
Health-related quality of life (HRQL) | 12 months
  The Pediatric Quality of Life Inventory (PedsQL) 4.0 is a 23-item generic HRQL scale not specific to pain. It is comprised of physical, emotional, social and school functioning subscales with each subscale containing 5 to 8 items. PedsQL4.0 is a reliable and valid measure of HRQL in AWC (Varni, Burwinkle, Katz, Meeske, & Dickinson, 2002). We will use age-appropriate versions of PedsQL4.0 (i.e., appropriate item wording for 12 and 13-18 year olds). Total and subscale scores will be used in analyses.
Self-efficacy | 12 months
  The Sherer's General Self-Efficacy Scale (GSES) is a 17-item scale that measures general belief in personal competence and has been used in children as young as 10 years old. Each item is scored on a 5-point Likert scale. Item scores are summed to provide an overall self-efficacy score to be used in analyses. The psychometric properties of the measure have been demonstrated in AWC (Hinds et al., 2000).
Healthcare utilization | 12 months
  Healthcare utilization related to pain will be examined as the number of visits/calls to primary care provider, emergency room visits, oncology clinic visits and hospitalizations (i.e., bed days of care). RN calls will not be included in healthcare utilization analyses. Data will be collected using adolescent self-report and medical health records (by site specific RAs at end of study).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stinson, RN, PhD, Principal Investigator — The Hospital for Sick Children

REFERENCES:
- [Result] Jibb LA, Cafazzo JA, Nathan PC, Seto E, Stevens BJ, Nguyen C, Stinson JN. Development of a mHealth Real-Time Pain Self-Management App for Adolescents With Cancer: An Iterative Usability Testing Study [Formula: see text]. J Pediatr Oncol Nurs. 2017 Jul/Aug;34(4):283-294. doi: 10.1177/1043454217697022. Epub 2017 Apr 4. PMID 28376666
- [Result] Jibb LA, Stevens BJ, Nathan PC, Seto E, Cafazzo JA, Johnston DL, Hum V, Stinson JN. Implementation and preliminary effectiveness of a real-time pain management smartphone app for adolescents with cancer: A multicenter pilot clinical study. Pediatr Blood Cancer. 2017 Oct;64(10). doi: 10.1002/pbc.26554. Epub 2017 Apr 19. PMID 28423223